CLINICAL TRIAL: NCT00566683
Title: Nurse-Administered Propofol Sedation by PCA Pump Versus Diazemuls / Pethidine in Outpatient Colonoscopy: A Randomized Controlled Study
Brief Title: Comparison Between Nurse-Administered Propofol Sedation and Diazemuls / Pethidine in Outpatient Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North District Hospital (Other)
Responsible Party: Poon Chi-Ming, North District Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CRE-2005.010-T
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2007-12-03 (Estimated); Status verified 2007-11

CONDITIONS: Colonoscopy
Keywords: Propofol; colonoscopy; sedation; pain; compare NAPS versus diazemuls in outpatient colonoscopy
MeSH Terms: conditions — Pain | interventions — Diazepam; Meperidine; Propofol; Alfentanil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Diazemuls-Pethidine
  Interventions: Drug: diazemuls, pethidine
- 2 (Active Comparator): Propofol- Alfentanil
  Interventions: Drug: Propofol and Alfentanil

INTERVENTIONS:
Drug: diazemuls, pethidine — 5mg Diazemuls and 25mg Pethidine one min. before procedure followed by bolus doses of 2.5mg Diazemuls / 12.5mg Pethidine at the discretion of endoscopists Maximal dose of 0.2mg/kg Diazemuls and 1mg/kg Pethidine
  Arms: 1
Drug: Propofol and Alfentanil — Loading dose of 40-60mg or 0.8mg/kg Propofol one min. before procedure Propofol 200mg + Alfentanil 0.5mg, 1.5ml per bolus (bolus dose of 14.3mg Propofol + 35ug Alfentanil) via PCA pump No maximal dose Zero lockout time
  Arms: 2

SUMMARY:
Colonoscopy is a common endoscopic procedure as an investigation of colorectal pathology. Different modalities of pain control have been described in the past. Propofol is a perfect drug for endoscopic procedure since it has the characteristic of fast onset, short half-life and early recovery. Its unfamiliarity and its potential cardiovascular and respiratory side effect make it unpopular to endoscopists. Recent reports showed propofol is safe in bolus titration by nurse in Caucasian in all endoscopic procedures. Our previous pilot study showed nurse administered propofol sedation (NAPS) is effective and safe and highly acceptable by Chinese patients. Here we conduct a randomized controlled study to compare the effectiveness of NAPS versus traditional sedation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 undergoing elective outpatient colonoscopy

Exclusion Criteria:

* American Society of Anesthesiologist Class III or above
* History of difficult endotracheal intubation
* Known allergy to propofol, eggs or soy products, opioid, benzodiazepines
* previous colectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2005-07; Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Pain | after recovery

SECONDARY OUTCOMES:
sedation | thorughout the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Ming Poon, MBBS, Principal Investigator — North District Hospital